CLINICAL TRIAL: NCT02467049
Title: ECG Versus Ultrasound-guided Positioning of the Peripherally Inserted Central Catheter (PICC) Tip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Study Nurse, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECG-PICC
Record Dates: First submitted 2015-05-26; First posted 2015-06-09 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Infection; Cancer; Malnutrition
Keywords: ECG; Ultrasound; Peripherally Inserted Central Catheters; PICC
MeSH Terms: conditions — Infections; Neoplasms; Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECG-guided insertion of PICC (Active Comparator): Placement of the PICC (Peripherally Inserted Central Catheter ) ECG-guided insertion.
  Interventions: Device: ECG-guided insertion of PICC; Device: ULTRASOUND-guided insertion of PICC
- ULTRASOUND-guided insertion of PICC (Experimental): Placement of the PICC (Peripherally Inserted Central Catheter ) ULTRASOUND-guided.
  Interventions: Device: ECG-guided insertion of PICC; Device: ULTRASOUND-guided insertion of PICC

INTERVENTIONS:
Device: ECG-guided insertion of PICC — Comparison of placement of a PICC (Peripherally Inserted Central Catheter) by ECG-guidance vs. ULTRASOUND-guidance
Device: ULTRASOUND-guided insertion of PICC — Comparison of placement of a PICC (Peripherally Inserted Central Catheter) by ECG-guidance vs. ULTRASOUND-guidance

SUMMARY:
In the prevention of thrombosis related to catheter placement it is important to have a right position of the catheter tip. Therefor we want to assess which technique is the most successful in the placing of a PICC.

DETAILED DESCRIPTION:
This is a randomised prospective single blinded study. All adult patients with an indication for PICC placement can be included. Patients will be randomised into two groups, one with ECG-guided placement followed by ultrasound control and the other with only ultrasound guided placement. After placement, in both groups, control radiography of the chest will be done which will be interpreted by an independent radiologist. For the ECG-guided group the ultrasound control of the tip position will be done by an independent, blind operator, after placement. For the only ultrasound guided placement group, the ultrasound will be done by a second operator during placement.

ELIGIBILITY:
Inclusion Criteria:

* All adults with indication for PICC

Exclusion Criteria:

* Age <18y
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with correct placement in the superior caval vein during PICC insertion, after either ECG or ultrasound guided insertion | Whitin 5 minutes after catheter-placement
  The aim of the study is a comparison between two techniques to control correct positioning of the PICC

SECONDARY OUTCOMES:
Duration of PICC-placement by ECG-guidance versus ultrasound-guidance | within 5 minutes
frequency of necessity of replacement after chest-x-ray control | 1 day
  PICC tip should be located in the superior caval vein, close to the entrance of the right atrium. Other locations lead to repositioning.

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Choustoulakis, MD, Principal Investigator — Department of Anaestesiology and Perioperative Medicine Acute and Chronic Pain Therapy.; Jan Poelaert, MD, PhD, Study Chair — Department of Anaestesiology and Perioperative Medicine Acute and Chronic Pain Therapy.; Matthias Raes, MD, Principal Investigator — Department of Anaestesiology and Perioperative Medicine Acute and Chronic Pain Therapy.
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No